CLINICAL TRIAL: NCT03786380
Title: Open-label Extension Study of Relamorelin for the Treatment of Diabetic Gastroparesis
Brief Title: Diabetic Gastroparesis Study 05
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Relamorelin program is being terminated solely based on a business decision.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3071-305-020; 2019-000406-30 (EudraCT Number)
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Results first posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-11

CONDITIONS: Gastroparesis
Keywords: Diabetic Gastroparesis
MeSH Terms: conditions — Gastroparesis | interventions — relamorelin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Relamorelin 10 μg (Experimental): Relamorelin 10 micrograms (μg) injected subcutaneously twice daily for up to approximately 22 months.
  Interventions: Drug: Relamorelin 10 μg

INTERVENTIONS:
Drug: Relamorelin 10 μg — Relamorelin 10 μg injected subcutaneously twice daily.

SUMMARY:
This open-label study is to assess the safety of continued treatment with relamorelin for participants who previously completed the RLM-MD-03 [NCT03420781] or RLM-MD-04 [NCT03383146] study and to provide treatment for these participants until relamorelin becomes commercially available or the Sponsor terminates development.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of either Study RLM-MD-03 or Study RLM-MD-04
* Ability to provide written informed consent (IC) prior to any study procedures and willingness and ability to comply with study procedures
* Demonstration of adequate compliance with the study procedures in Study RLM-MD-03 or RLM-MD-04, in the opinion of the investigator.

Exclusion Criteria:

* Participant is planning to receive an investigational drug (other than study intervention) or investigational device at any time during Study 3071-305-020
* Participant has an unresolved adverse event (AE) from a lead-in study, ie, a clinically significant finding on physical examination, clinical laboratory test, or 12-lead electrocardiogram (ECG) that, in the investigator's opinion, would limit the participant's ability to participate in or complete the study
* Any other reason that, in the investigator's opinion, would confound proper interpretation of the study or expose a participant to unacceptable risk, including renal, hepatic, or cardiopulmonary disease
* Females who are pregnant, nursing, or planning a pregnancy during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2020-10-05 (Actual); Study Completion 2020-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harvy Schneier, Study Director — Allergan
Locations (486):
- United States (189):
  - Pinnacle Research Group, Anniston, Alabama
  - North Alabama Research Center, LLC, Athens, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Digestive Health Specialist of the South East, Dothan, Alabama
  - G & L Research, LLC, Foley, Alabama
  - Alabama Medical Group, PC, Mobile, Alabama
  - Del Sol Research Management, LLC, Chandler, Arizona
  - Phoenix Clinical LLC., Phoenix, Arizona
  - Adobe Clinical Research LLC, Tucson, Arizona
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Preferred Clinical Research Partners, Little Rock, Arkansas
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - Arkansas Gastroenterology, North Little Rock, Arkansas
  - HCP Clinical Research LLC, Anaheim, California
  - Hope Clinical Research, Canoga Park, California
  - GW Research Inc, Chula Vista, California
  - Kindred Medical Institute for Clinical Trials, LLC, Corona, California
  - Aurora Care Clinic, LLC, Costa Mesa, California
  - Diagnamics Inc., Encinitas, California
  - Valley View Wellness and Medical Center - VVCRD Clinical Research, Garden Grove, California
  - University of California San Diego, La Jolla, California
  - Om Research LLC, Lancaster, California
  - Torrance Clinical Research Institute, Inc., Lomita, California
  - Tibor Rubin VA Medical Center, Long Beach, California
  - Angel City Research Inc., Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Stanford Hospital, Palo Alto, California
  - TriWest Research Associates, Poway, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Medical Associates Research Group, Inc, San Diego, California
  - Syrentis Clinical Research, Santa Ana, California
  - Upland Clinical Research, Upland, California
  - New Hope Research Development, Whittier, California
  - University of Colorado, Denver, Aurora, Colorado
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Denver Esophageal and Stomach Center, Englewood, Colorado
  - Gastroenterology Associates of Fairfield County, P.C., Bridgeport, Connecticut
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Visionary Investigators Network, Aventura, Florida
  - Gastro Florida, Clearwater, Florida
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of West Florida, Clearwater, Florida
  - ALL Medical Research LLC, Cooper City, Florida
  - American Research Institute, Inc, Cutler Bay, Florida
  - Top Medical Research, Cutler Bay, Florida
  - Palmetto Research, LLC, Hialeah, Florida
  - Vida Clinical Trials, Homestead, Florida
  - Nature Coast Clinical Research, Inverness, Florida
  - University of Florida, Jacksonville, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Cfagi Llc, Maitland, Florida
  - APF Research LLC, Miami, Florida
  - AMPM Research Clinic, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Florida Research Center, Inc., Miami, Florida
  - Panax Clinical Research, Miami Lakes, Florida
  - Savin Medical Group LLC, Miami Lakes, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Sensible Healthcare, Ocoee, Florida
  - Gulf Region Clinical Research Institute, Pensacola, Florida
  - University of South Florida, Tampa, Florida
  - Gastro Florida, Tampa, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - Atlanta Diabetes Associates, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - River Birch Research Alliance, LLC, Blue Ridge, Georgia
  - Gwinnett Research Institute, Buford, Georgia
  - Summit Clinical Research, LLC., Carnesville, Georgia
  - iResearch Atlanta LLC, Decatur, Georgia
  - Infinite Clinical Trials, Riverdale, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center, PA, Idaho Falls, Idaho
  - North Shore University Health System, Evanston, Illinois
  - Southwest Gastroenterology, Oak Lawn, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - American Research, LLC, Jeffersonville, Indiana
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - Integrated Clinical Trial Services Inc, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Health Science Research Center, Pratt, Kansas
  - Cotton-O'Neil Clinical Research Center - Digestive Health, Topeka, Kansas
  - Professional Research Network of Kansas, LLC, Wichita, Kansas
  - Via Christi Clinic, PA, Wichita, Kansas
  - Tri-State Gastroenterology, Crestview Hills, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Delta Research Partners, Bastrop, Louisiana
  - Avant Research Associates LLC, Crowley, Louisiana
  - Cronola LLC, Houma, Louisiana
  - Centex Studies, Inc. - Lake Charles- Clinical Trials of SWLA, LLC, Lake Charles, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - New Orleans Research Institute - Metropolitan Gastroenterology Associates, Metairie, Louisiana
  - Clinical Trials of America, Inc., West Monroe, Louisiana
  - Metropolitan Gastroenterology Group PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Gastro Center of Maryland, Columbia, Maryland
  - Woodholme Gastroenterology Associates, P.A., Glen Burnie, Maryland
  - Commonwealth Clinical Studies, PLLC., Brockton, Massachusetts
  - Coastal Research Associates, Inc., South Weymouth, Massachusetts
  - Boston VA Healthcare System, West Roxbury, Massachusetts
  - Biocon Clinical Research, LLC, Caro, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Aa Mrc, Llc, Flint, Michigan
  - National Clinical, LLC, Hamtramck, Michigan
  - Henry Ford Health System, Novi, Michigan
  - Troy Gastroenterology, PC dba Center for Digestive Health, Troy, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - MNGI Digestive Health, Coon Rapids, Minnesota
  - Washington University in St. Louis, St Louis, Missouri
  - Montana Medical Research, Missoula, Montana
  - Heartland Clinical Research, Inc, Omaha, Nebraska
  - Clinical Research of South Nevada, Las Vegas, Nevada
  - Advanced Biomedical Research of America, Las Vegas, Nevada
  - Digestive Disease Specialists, Las Vegas, Nevada
  - Palm Research Center, Las Vegas, Nevada
  - Test Center 3, Brick, New Jersey
  - AGA Clinical Research Associates, LLC, Egg Harbor, New Jersey
  - Lovelace Scientific Resources, Inc., Albuquerque, New Mexico
  - Long Island Gastrointestinal Research Group LLP, Great Neck, New York
  - Queens Hospital Center, Jamaica, New York
  - United Health Services Hospitals, Inc., Johnson City, New York
  - NYU Winthrop Hospital, Clinical Trials Center, Mineola, New York
  - Weill Cornell Medical College, New York, New York
  - Asheville Gastroenterology Associates, Asheville, North Carolina
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Test Center 2, Charlotte, North Carolina
  - PMG Research of Charlotte, LLC, Concord, North Carolina
  - Carolina Digestive Health Associates, PA, Davidson, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Triad Clinical Trials, Greensboro, North Carolina
  - Vidant Multispeciality Clinic - Kinston, Kinston, North Carolina
  - Diabetes and Endocrinology Consultants, PC, Morehead City, North Carolina
  - PMG Research Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Dayton Gastroenterology,Inc., Beavercreek, Ohio
  - The MetroHealth System MHS, Cleveland, Ohio
  - Digestive Disease & Surgery Institute, Cleveland, Ohio
  - Endocrinology Research Associates, Inc., Columbus, Ohio
  - The Ohio State University, Wexner Medical Center, Columbus, Ohio
  - Aventiv Research, Inc., Columbus, Ohio
  - Hometown Urgent Care and Research, Columbus, Ohio
  - Clinical Inquest Center Ltd., Dayton, Ohio
  - Family Practice Center of Wadsworth, Inc. DBA New Venture Medical Research, Wadsworth, Ohio
  - Digestive Disease Specialists Inc, Oklahoma City, Oklahoma
  - Memorial Clinical Research, Oklahoma City, Oklahoma
  - Options Health Research, LLC, Tulsa, Oklahoma
  - Family Medical Associates, Research Department, Levittown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Guthrie Clinical Research, Sayre, Pennsylvania
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Montgomery Medical, Inc., Smithfield, Pennsylvania
  - Preferred Primary Care Physicians, Jacob Murphy, Uniontown, Pennsylvania
  - Partners in Clinical Research, LLC, Cumberland, Rhode Island
  - Clinical Trials of South Carolina, Charleston, South Carolina
  - Gastroenterology Associates, PA, Greenville, South Carolina
  - Health Concepts, Rapid City, South Dakota
  - Clinsearch, Chattanooga, Tennessee
  - Gastro One, Germantown, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Clinical Research Institute, LLC, Arlington, Texas
  - Avant Research Associates,LLC, Austin, Texas
  - DiscoveResearch, Inc., Beaumont, Texas
  - ClinRx Research, LLC, Carrollton, Texas
  - Texas Tech University Health Sciences, Center Division of Gastroenterology, El Paso, Texas
  - DHAT Research Institute, Garland, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Biopharma Informatic Inc., Research Center, Houston, Texas
  - Rodriguez Clinical Trials, Houston, Texas
  - Amir Ali Hassan, MD, PA, Houston, Texas
  - Digestive Center of South Texas, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - SAGACT PLLC., San Antonio Gastroenterology Associates, PA, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Advanced Research Institute, Inc., Ogden, Utah
  - Test Center, Salt Lake City, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Verity Research Inc., Fairfax, Virginia
  - Blue Ridge Medical Research, Lynchburg, Virginia
  - Manassas Clinical Research Centre, Manassas, Virginia
  - VA Medical Center McGuire VAMC, Richmond, Virginia
  - Test Center 4, Roanoke, Virginia
  - Cardinal Internal Medicine, Woodbridge, Virginia
  - Washington Gastroenterology PLLC, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia
- Argentina (6):
  - Maffei Centro Medico-Investigacion Clinica Aplicada, C.a.b.a., Buenos Aires
  - Hospital Sirio Libanes, CABA, Buenos Aires
  - CIPREC, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas de Rosario, Rosario, Santa Fe Province
  - Instituto de hematología y medicina clínica "Dr. Rubén Dávoli", Rosario, Santa Fe Province
  - Centro Universitario de Investigacion en Farmacologia Clinic, Corrientes
- Australia (5):
  - Nepean Hospital, Kingswood, New South Wales
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital - Central Adelaide Local Health Network Incorporated, Adelaide, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Austria (8):
  - Ordination, Saint Stefan, Styria
  - Medizinische Universitaet Innsbruck, Innsbruck, Tyrol
  - VIVIT Institute, am LKH Feldkirch, Feldkirch, Vorarlberg
  - Klinikum Klagenfurt am Wörthersee, Klagenfurt
  - Privatklinik Wehrle-Diakonissen, Salzburg
  - Oö. Gesundheits- und Spitals-AG/LKH Steyr, Steyr
  - Krankenanstalt Rudolfstiftung Wien, Vienna
  - KH Hietzing, Vienna
- Belgium (5):
  - AZ Sint Lucas Brugge, Bruges, Antwerpen
  - Universitair Ziekenhuis Antwerpen, Gastro-Enterologie,, Edegem, Antwerpen
  - Hôpitaux Iris Sud - Joseph Bracops, Brussels
  - UZ Brussel, Jette
  - CHC - Clinique Saint-Joseph, Liège
- Brazil (14):
  - Hospital Universitário Walter Cantídio, Fortaleza, Ceará
  - Centro de Pesquisa Clinica do Brasil, Brasília, Federal District
  - Quanta Diagnóstico e Terapia, Curitiba, Paraná
  - Hospital Universitário João de Barros Barreto - UFPA, Belém, Pará
  - Hospital Sao Vicente de Paulo, Passo Fundo- RS, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUC-RS, Porto Alegre, Rio Grande do Sul
  - Instituto Catarinense de Endocrinologia e Diabetes (ICED), Joinville, Santa Catarina
  - Scentryphar Pesquisa Clínica Ltda, Campinas, São Paulo
  - Instituto de Pesquisa Clínica em Campinas, Campinas, São Paulo
  - Universidade de Sao Paulo (USP) - Hospital das Clinicas da F, Cerqueira Cesar - Sao Paulo, São Paulo
  - IPEC-Instituto de Pesquisa Clinica, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica Ltda, São Paulo, São Paulo
  - Instituto de Estudos e Pesquisas Clínicas do Ceará - IEP/CE - Oncology, Fortaleza
- Bulgaria (6):
  - MHAT Yuliya Vrevska Byala, Byala
  - MHAT Dobrich AD, Dobrich
  - MHAT Dr. Tota Venkova AD, Gabrovo
  - UMHAT - Kaspela- EOOD, Plovdiv
  - Medical Center Asklepion - Humane Medicine Research EOOD, Sofia
  - Alexandrovska University Hospital, Sofia
- Canada (15):
  - University of Calgary, Calgary, Alberta
  - Alberta Diabetes Institute, Edmonton, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Eastern Health, St. John's, Newfoundland and Labrador
  - South Shore Medical Arts, Bridgewater, Nova Scotia
  - Dr. Anil K. Gupta Medicine Professional Corporation, Etobicoke, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Science Centre, Toronto, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - Toronto Liver Centre, Toronto, Ontario
  - CISSS de la Monteregie-Centre, Greenfield Park, Quebec
  - Recherche GCP Research, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal - CHUM, Montreal, Quebec
  - Central Alberta Research Centre, Red Deer
  - Toronto Digestive Disease Associates, Vaughan
- Colombia (8):
  - Rodrigo Botero S.A.S., Medellín, Antioquia
  - Centro Cardiovascular y de Diabetes, Barranquilla, Atlántico
  - Fundación BIOS, Barranquilla, Atlántico
  - Endocare Ltda., Bogota, Cundinamarca
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Medplus Medicina Prepagada, Bogotá, Distrito Capltal
  - Centro Medico Imbanaco de Cali S.A., Cali, Distrito Capltal
  - IPS Centro Medico Julian Coronel S.A, Cali, Valle del Cauca Department
- Denmark (5):
  - Gastroenheden, Hvidovre hospital, Hvidovre, Kobenhavn
  - Aalborg University Hospital, Aalborg
  - Steno Diabetes Center Copenhagen, Hellerup
  - Nordsjaellands Hospital, Hilleroed
  - MEA KFA, Aarhus, Århus
- France (10):
  - CHU de Bordeaux - Hôpital Haut-Lévêque, Pessac, Gironde
  - Hôpital Louis-Mourier, Colombes
  - Corbeil Essonnes, Corbeil-Essonnes
  - Service d'hépato-gastroentérologie - 7°D, Grenoble
  - Hospices Civils de Lyon - Hôpital Edouard Herrriot, Lyon
  - CHU Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - Hopital Charles Nicolle, Rouen
  - CHRU Nancy, Vandœuvre-lès-Nancy
  - Centre de Recherche Clinique, Vénissieux
- Germany (12):
  - Klinische Forschung Karlsruhe GmbH, Karlsruhe, Baden-Wurttemberg
  - Praxis Dr. Etzrodt-Walter und Kollegen, Ulm, Baden-Wurttemberg
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Diabetologische Schwerpunktpraxis, Bad Berleburg, North Rhine-Westphalia
  - Klinische Forschung Dresden GmbH, Dresden, Saxony
  - Studienzentrum Schwittay, Böhlen
  - Universitätsklinikum Giessen und Marburg GmbH, Giessen
  - Klinische Forschung Hamburg GmbH, Hamburg
  - Clinical Research Hamburg GmbH, Hamburg
  - Israelitisches Krankenhaus, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - KRH Klinikum Siloah, Hanover
- Hungary (7):
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger, Heves County
  - Coromed SMO, Pécs, Pécs
  - First Department of Medicine, University of Szeged, Szeged, Szaged
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg, Zala County
  - Semmelweis University, Budapest
  - Stra¡zshegy Medicina, Budapest
  - Hetenyi Geza Hospital, Szolnok
- India (30):
  - King George Hospital, Visakhapatnam, Andhra Pradesh
  - Dr. Jivraj Mehta Smarak Health Foundation Bakeri Medical Res, Ahmedabad, Gujarat
  - Zydus Hospital, Ahmedabad, Gujarat
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Lifecare Clinic and Research Centre - Internal Med/Diabetolo, Bangalore, Karnataka
  - Diacon Hospital and research Center, Bengaluru, Karnataka
  - Victoria Hospital Bangalore Medical College and Research Ins, Bengaluru, Karnataka
  - Rajalakshmi Hospital, Bengaluru, Karnataka
  - Vinaya Hospital & Research Centre, Mangalore, Karnataka
  - Chopda Medicare & Research Centre Pvt.Ltd, Magnum Heart Institute, Nashik, Maharashtra
  - B. J. Government Medical College and Sassoon General Hospitals, Pune, Maharashtra
  - Grant Medical Foundation Ruby Hall Clinic, Pune, Maharashtra
  - University Hospital, Pune, Maharashtra
  - Noble Hospital, Pune, Maharashtra
  - S.P.Medical College & Group of Hospitals Bikaner, Bikaner, Rajasthan
  - S.R. Kalla Memorial Gastro and General Hospital, Jaipur, Rajasthan
  - Sawai Man Singh Hospital, Jaipur, Rajasthan
  - Sir Ganga Ram Hospital (SGRH), Jaipur, Rajasthan
  - Marudhar Hospital, Jaipur, Rajasthan
  - Eternal Hospital, Unit of Eternal Heart Care Centre and Research Institute Pvt. Ltd., Jaipur, Rajasthan
  - Madras Medical College & Rajiv Gandhi Govt. General Hospital, Chennai, Tamil Nadu
  - M.V. Hospital for Diabetes & Diabetes Research Centre, Chennai, Tamil Nadu
  - Kovai Diabetes Speciality Centre, Coimbatore, Tamil Nadu
  - Arthur Asirvatham Hospital, Madurai, Tamil Nadu
  - M V Hospital & Research Centre, Lucknow, Uttar Pradesh
  - IPGME&R and SSKM Hospital, Kolkata, West Bengal
  - M. S. Ramaiah medical College and Hospitals - Gastroenterolo, Bangalore
  - Gleneagles Global Hospital, Hyderabad
  - Kumudini Devi Diabetes Research Center, Hyderabad
  - Bhatia Hospital, Mumbai
- Israel (7):
  - Soroka University Medical Center, Beersheba
  - Bnai Zion M.C., Haifa
  - E. Wolfson Medical Center, Holon
  - Digestive Diseases Institute, Jerusalem
  - Gastroenterology Institute, Petah Tikva
  - Endocrinology & Diabetes Center, Safed
  - Gastroenterology Institute, Tel Aviv
- Italy (15):
  - IRCCS Policlinico San Donato, San Donato Milanese, Milan
  - Clinical Institute Beato Matteo, Vigevano, Pavia
  - Policlinico Gemelli, Divisione di Endocrinologia e Malattie del Metabolismo, Rome, Rome Roma
  - Ospedale Cardinal Massaia, Asti
  - University of Bari, Bari
  - Azienda Ospedaliera Rilievo Nazionale Alta Specialita (ARNAS) Garibaldi, Catania
  - Universita Magna Graecia di Catanzaro, Catanzaro
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - Universita degli Studi di Napoli Federico II, Napoli
  - Azienda Opsedaliera di Padova, Padua
  - IRCCS S.Matteo Hospital Foundation, University of Pavia, Pavia
  - University of Pisa - Cisanello Hospital, Pisa
  - Gruppo Humanitas - Humanitas Research Hospital, Rozzano
  - Universita' Di Salerno- Aou Ruggi D'aragona, Salerno
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
- Latvia (4):
  - Polana-D, Daugavpils
  - Ogorelova Jelena GP, Krāslava
  - Pauls Stradins Clinical University Hospital, Endokrinologijas nodala, Riga
  - Digestive Diseases Centre GASTRO, Riga
- Malaysia (4):
  - Hospital Sultanah Bahiyah, Alor Star, Kedah
  - University Malaya Medical Centre, Kuala Lumpur
  - Universiti Sains Malaysia, Kubang Kerian
  - Hospital Taiping, Taiping
- Mexico (20):
  - Centro de Investigacion Morales Vargas - CIMOVA, León, Guanajuato
  - Centro de Diabetes de Pachuca, Pachuca, Hidalgo
  - Unidad de Investigación Clínica Cardiometabolica de Occidente, Guadalajara, Jalisco
  - Consultorio Medico, Guadalajara, Jalisco
  - Unidad de Investigación clínica y atención Médica HEPA S.C., Guadalajara, Jalisco
  - Clinicos Asociados BOCM SC, Mexico City, Mexico City
  - Clinica OMEGA, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion, Mexico City, Mexico City
  - Medical and Nutritional Trials, México DF, Mexico City
  - Instituto de Diabetes Obesidad y Nutrición SC, Cuautla, Morelos
  - Accelerium Clinical Research, Monterrey, Nuevo León
  - Centro Medico Christus Muguerza Sur, Monterrey, Nuevo León
  - Investigación Médica Sonora, S.C., Hermosillo, Sonora
  - Centro Especializado en Investigación Clínica S.C., Boca del Rio, Veracruz
  - Centro de Desarrollo Biomédico, Mérida, Yucatán
  - Practice Dr Gerardo Gonzalez, Acapulco
  - Hospital Cardiológica Aguascalientes, Aguascalientes
  - Dioderm Instituto de Investigación, Durango
  - CIADEN (Centro de Investigación y Atención de Diabetes, Endocrinología y Nutrición), Durango
  - Sociedad de Metabolismo y Corazón, S.C., Veracruz
- Philippines (7):
  - Perpetual Succor Hospital, Cebu City
  - West Visayas State University Medical Center, Iloilo City
  - Ospital ng Makati, Makati City
  - Manila Doctors Hospital, Manila
  - San Juan De Dios Educational Foundation, Inc., Pasay
  - St. Luke's Medical Center, Quezon City
  - Cardinal Santos Medical Center, San Juan City
- Poland (16):
  - NZOZ Vita - Diabetica Malgorzata Buraczyk, Diabetes Clinic,, Bialystok, Bia|ystok
  - Centrum Medyczne Pratia Warszawa, Warsaw, Warazawa
  - Szpital Uniwestytetu Medycznego w Bialymstoku, Bialystok
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Vitamed, Bydgoszcz
  - Centrum Medyczne Lukamed, Chojnice
  - Silmedic Sp z o o, Katowice
  - Specjalistyczny Gabinet Neurologiczny Marta Banach, Krakow
  - CenterMed Krakow Ltd, Krakow
  - Centrum Medyczne Medyk, Lublin
  - Wojewodzki Szpital Specjalistyczny w Olsztynie, Olsztyn
  - Oddzial Gastroenterologii Mazowieckie Centrum Rehabilitacji Stocer sp. Z o.o., Pruszków
  - Endoskopia SP. Z O.O., Sopot
  - Powiatowe Centrum Medyczne w Wołowie, Wołów
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroclaw
  - Zamość, Zamość
- Romania (5):
  - Sana Medical Center, Bucharest
  - National Institute of Endocrinology, Bucharest
  - AMES Research Center SRL, Călăraşi
  - ClinTrial Medical Center, Pulmonology Department, Dobrosloveni Resca, Olt County
  - Polisano-Clinic, Sibiu
- Russia (12):
  - Scientific Institute of Clinical and Experimental Lymphology, Novosibirsk, Novosibirsk Oblast
  - North-Western State Medical University named after I. I. Mechnikov, Saint Petersburg, Sankt-Peterburg
  - Millitary-medical Academy, department of hospital therapy, Saint Petersburg, Sankt-Peterburg
  - Kazan State Medical University, Kazan'
  - Saint-Petersburg City Pokrovskaya Hospital, Leningrad Region
  - FSBI National medical endocrinology research centre, Moscow
  - Moscow Regional Research Clinical Institute named by MF Vladimirski, Moscow
  - Nizhegorodsky Regional Clinical Hospital named after N. A. Semashko, Nizhny
  - Rostov on Don, Rostov-on-Don
  - Rostov State Medical University, Rostov-on-Don
  - MUZ City Clinical Hospital 9, Saratov
  - Saratov City Clinical Hospital 12, Saratov
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Changi General Hospital, Singapore
- South Africa (9):
  - FARMOVS, Bloemfontein, Free State
  - Soweto CTC, Johannesburg, Gauteng
  - Wits Clinical Research, Johannesburg, Gauteng
  - Synexus Stanza Clincal Reaserch Centre, Pretoria, Gauteng
  - Endocare Research, Paarl, Western Cape
  - Synexus Helderberg Clinical Research Centre, Cape Town
  - TREAD Research, Cape Town
  - Syenxus Watermeyer Dedicated Research, Val de Grace
  - Moriana Clinical Research, Winnie Mandela
- South Korea (3):
  - Chonbuk National University Hospital, Jeonju, Jeollabuk-do
  - Sanggye Paik Hospital, Inje University College of Medicine, Seoul
  - Asan Medical Center, Seoul
- Spain (7):
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Principe de Asturias, Madrid
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario Miguel Servet, Zaragoza
- Thailand (3):
  - Phramongkutklao Hospital, Bangkok
  - Faculty of Medicine, Siriraj Hospital, Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- Ukraine (33):
  - State Institution Ukrainian State Research Institute, Dnipro, Dnipropetrovsk Oblast
  - "Kryvyi Rih City Hospital #3" of Dnipropetrovsk Regional Council, Dnipropetrovsk Region, Dnipropetrovsk Oblast
  - Ivano-Frankivsk National Medical University, Ivano-Frankivsk, Ivano-Frankivsk Oblast
  - Kyiv city clinical endocrinology center, department of general endocrine pathology and metabolism, c. Kyiv, Kyiv, Kyïv
  - DRRI-Vinnytsia National Pirogov Memorial Medical University, Vinnytsia, Vinnytsia Oblast
  - Municipal Institution Lutsk City Clinical Hospital, Lutsk, Volyos'ka Oblast'
  - Municipal nonprofit entity "Chernigiv city hospital #2" of Chernigiv municipal council, therapeutic department, Chernihiv
  - Regional municipal institution "Chernivtsi's regional clinical hospital", gastroenterological department, Higher state educational establishment of Ukraine "Bukovinian state medical university", department of internal medicine and infectious diseases, c.C, Chernivtsi
  - Regional Public Organization Chernivtsi Regional Endocrinology Center, Chernivtsi
  - SU Clinic of medical academy of SI Dnepropetrovsk medical cacadamy of MoH of Ukraine, Dnipro
  - Ivano-Frankivsk Central City Clinical Hospital, Ivano-Frankivsk
  - Municipal nonprofit entity "City clinical hospital #2 n.a. Prof.O.O.Shalimov" of Kharkiv municipal council, department of endocrinology, Kharkiv
  - "State Institution "National Institute of Therapy named after. L.T. Maloi NAMNU" / Government Institution "L.T.Malaya Therapy National Institute of the National Academy of Medical Sciences of Ukraine", Department of the study of diseases of the digestive, Kharkiv
  - Clinical Endocrinology of SI V.Danilevsky Institute for endocrine pathology problems National Academy of Medical sciences of Ukraine, Kharkiv
  - Communal Institution Kherson City Clinical Hospital, Kherson
  - Limited Liability Company "Medical and Diagnostic Center "ADONIS Plus", outpatient department, c. Kyiv, Kyiv
  - Kyiv Railway Clinical Hospital #2 of Branch Healthcare Center of the PJSC Ukranian Railway, Endocrynology Department, Kyiv
  - Medical Center Universal Clinic OberigMedical Center Universal Clinic Oberig / Medical Center "Universal Clininc "Oberig" of LLC "Capital", Gastroenterological Center, c. Kyiv, Kyiv
  - Polyclinic of medical services and rehabilitation department of State Joint-Stock Holding Company Artem, day-patient unit, Kyiv
  - Institute of Endocrinology and Metabolism im. V. P. Komisarenka NAMS Ukraine, Kyiv
  - City Hospital #1, department of endocrinology, c. Mykolayiv, Mykolaiv
  - Odessa Railway Clinical Hospital of Branch of HC JSC Ukrzaliznytsia, Odessa National Medical University, Odesa
  - Communal Institution "Odesa Regional Clinical Hospital", Out-patient department, Odesa
  - Poltava Regional Clinical Hospital, Poltava
  - Municipal Institution of Sumy Regional Council Sumy Regional Clinical Hospital, Sumy
  - Ternopil University Hospital, Regional Center for Gastroenterology with Hepatology, Department of Gastroenterology, Ternopil
  - Private Small-Scale Enterprise Medical Center Pulse, Vinnytsia
  - Medical Center of the Limited Liability Company "Health Clinic", Medical Clinical Research Center, Department of Gastroenterology, Hepatology and Endocrinology, Vinnytsia
  - Vinnytsia Regional Clinical highly specialized Endocrinology Centre, Vinnytsia
  - Municipal nonprofit entity "Vinnytsia's city clinical hospital #1", gastroenterological department, Vinnytsia National Pirogov Memorial Medical University, department of propedeutics of internal medicine, c. Vinnytsia, Vinnytsia
  - 6th City Clinical Hospital, c. Zaporizhzhia, Zaporizhzhia
  - "Municipal Institution ""City Hospital #7"", polyclinic department, c. Zaporizhzhia", Zaporizhzhia
  - Municipal Institution-Zaporizhzhia Regional Clinical Hospital, Zaporizhzhia
- United Kingdom (18):
  - Royal Oldham Hospital, Oldham, Lancashire
  - MAC Research, Exchange House, Cannock, Staffordshire
  - University Hospitals of North Midlands, Stoke-on-Trent, Staffordshire
  - MAC Research, Barnsley
  - MAC Clinical Research, Kaman Court, Blackpool
  - Mid Essex Hospital Services NHS Trust Broomfield Hospital, Chelmsford
  - Western General Hospital Edinburgh, Edinburgh
  - MAC Clinical Research, Monarch House, Leeds
  - MAC Clinical Research, Liverpool
  - Wingate Institute, London
  - University College London Hospita, London
  - MAC Clinical Research Manchester, Manchester
  - University Hospital of South Manchester, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Biomedical Research Centre, Nottingham
  - MAC Clinical Research, GAC House, Stockton-on-Tees
  - St George's Hospital, Tooting
  - Royal Wolverhampton NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who completed relamorelin studies: RLM-MD-03 [NCT03420781] and RLM-MD-04 [NCT03383146] were eligible to enroll in this open-label safety study.
Groups:
- Relamorelin/Relamorelin/Relamorelin: Relamorelin 10 micrograms (μg) injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received relamorelin 10 μg in the 40-week placebo-controlled treatment period and relamorelin 10 μg in the 6-week randomized withdrawal period (RWP) of RLM-MD-03.
- Relamorelin/Placebo/Relamorelin: Relamorelin 10 μg injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received relamorelin 10 μg in the 40-week placebo-controlled treatment period and placebo-matching relamorelin in the 6-week RWP of RLM-MD-03.
- Placebo/Relamorelin/Relamorelin: Relamorelin 10 μg injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received placebo-matching relamorelin in the 40-week placebo-controlled treatment period and relamorelin 10 μg in the 6-week RWP of RLM-MD-03.
- Relamorelin/Relamorelin: Relamorelin 10 μg injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received relamorelin 10 μg in double-blind treatment period of RLM-MD-04 for up to 52 weeks.
- Placebo/Relamorelin: Relamorelin 10 μg injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received placebo-matching relamorelin in the double-blind treatment period of RLM-MD-04 for up to 52 weeks.
Period: Overall Study
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
Started | 35 | 22 | 54 | 63 | 28
Safety Population (Safety Population included all participants who received ≥1 administration of study treatment.) | 35 | 22 | 54 | 62 | 28
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 35 | 22 | 54 | 63 | 28
Not completed — Adverse Event | 1 | 0 | 0 | 3 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2 | 2 | 1 | 2
Not completed — Lost to Follow-up | 3 | 0 | 1 | 2 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0
Not completed — Study Terminated by the Sponsor | 30 | 20 | 50 | 57 | 23
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Population included all participants enrolled in the study.
Groups:
- Relamorelin/Relamorelin/Relamorelin: Relamorelin 10 μg injected subcutaneously twice daily for up to approximately 22 months in this study. Participants in this arm group received relamorelin 10 μg in the 40-week placebo-controlled treatment period and relamorelin 10 μg in the 6-week RWP of RLM-MD-03.
- Total: Total of all reporting groups
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin | Total
Number analyzed (Participants) | 35 | 22 | 54 | 63 | 28 | 202
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.60) | 63.4 (11.87) | 55.7 (10.36) | 57.3 (9.19) | 58.5 (10.44) | 58.1 (10.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 14 | 38 | 46 | 22 | 146
  Male | 9 | 8 | 16 | 17 | 6 | 56
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 8 | 25 | 16 | 6 | 70
  Not Hispanic or Latino | 20 | 14 | 29 | 47 | 22 | 132
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 0 | 0 | 0 | 3
  Asian | 0 | 0 | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 11 | 13 | 8 | 37
  White | 31 | 18 | 43 | 48 | 20 | 160
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced One or More Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE is an AE that begins or worsens after receiving study drug.
Time Frame: Up to approximately 22 months
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
Number analyzed (Participants) | 35 | 22 | 54 | 62 | 28
Participants | 16 | 11 | 27 | 27 | 16

2. Primary Outcome: Number of Participants With Potential Clinically Significant (PCS) Clinical Laboratory Results
Description: Clinical Laboratory tests included hematology, chemistry and urinalysis tests. The investigator determined if the results were clinically significant. Only those categories where at least 1 person had a non-PCS value at Baseline and met the PCS criterion at least once during postbaseline are reported.
Time Frame: Baseline (Day 1) up to approximately 22 months
Population: Safety Population included all participants who received ≥1 administration of study treatment. Number analyzed is the number of participants with non-PCS baseline values and at least one post-baseline assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
Number analyzed (Participants) | 35 | 22 | 54 | 62 | 28
Participants
  Eosinophils Absolute Cell Count [10^9/liter (L)]: >3×Upper Limit of Normal Value (ULN): number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Eosinophils Absolute Cell Count [10^9/liter (L)]: >3×Upper Limit of Normal Value (ULN) | 0 | 1 | 0 | 0 | 0
  Hematocrit (RATIO): >1.1×ULN: number analyzed (Participants) | 34 | 21 | 50 | 61 | 28
  Hematocrit (RATIO): >1.1×ULN | 0 | 0 | 1 | 1 | 0
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN): number analyzed (Participants) | 34 | 21 | 50 | 61 | 28
  Hematocrit (RATIO): <0.9×Lower Limit of Normal Value (LLN) | 1 | 1 | 3 | 3 | 1
  Hemoglobin [grams (g)/L]: <0.9×LLN: number analyzed (Participants) | 34 | 21 | 51 | 60 | 28
  Hemoglobin [grams (g)/L]: <0.9×LLN | 2 | 5 | 11 | 3 | 2
  Lymphocytes Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 33 | 22 | 53 | 60 | 27
  Lymphocytes Absolute Cell Count (10^9/L): >1.5×ULN | 0 | 0 | 0 | 1 | 0
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 33 | 22 | 53 | 60 | 27
  Lymphocytes Absolute Cell Count (10^9/L): <0.8×LLN | 0 | 1 | 0 | 1 | 0
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN: number analyzed (Participants) | 34 | 22 | 52 | 59 | 28
  Mean Corpuscular Volume [femtoliter(fL)]: >1.1×ULN | 0 | 0 | 1 | 0 | 0
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN: number analyzed (Participants) | 32 | 21 | 52 | 61 | 28
  Neutrophils Absolute Cell Count (10^9/L): >1.5×ULN | 1 | 1 | 1 | 0 | 0
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN: number analyzed (Participants) | 32 | 21 | 52 | 61 | 28
  Neutrophils Absolute Cell Count (10^9/L): <0.8×LLN | 1 | 1 | 0 | 0 | 0
  Red Blood Cell Count (10^12/L): <0.9×LLN: number analyzed (Participants) | 34 | 21 | 53 | 60 | 28
  Red Blood Cell Count (10^12/L): <0.9×LLN | 1 | 2 | 4 | 0 | 0
  White Blood Cell Count (10^9/L): <0.7×LLN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  White Blood Cell Count (10^9/L): <0.7×LLN | 0 | 0 | 0 | 0 | 1
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Alanine Aminotransferase [Serum Glutamic Pyruvic Transaminase (SGPT)] [unit(U)/L]: >=3×ULN | 1 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Aspartate Aminotransferase [Serum Glutamic Oxaloacetic Transaminase (SGOT)] (U/L): >=3×ULN | 1 | 1 | 0 | 0 | 0
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN: number analyzed (Participants) | 34 | 20 | 53 | 61 | 28
  Bicarbonate (HCO3) [millimoles (mmol)/L]: >1.1×ULN | 1 | 0 | 1 | 0 | 0
  Bicarbonate (HCO3) (mmol/L): <0.9×LLN: number analyzed (Participants) | 34 | 20 | 53 | 61 | 28
  Bicarbonate (HCO3) (mmol/L): <0.9×LLN | 1 | 0 | 1 | 1 | 1
  Blood Urea Nitrogen (mmol/L): >1.2×ULN: number analyzed (Participants) | 29 | 19 | 51 | 60 | 26
  Blood Urea Nitrogen (mmol/L): >1.2×ULN | 7 | 3 | 10 | 4 | 2
  Calcium (mmol/L): >1.1×ULN: number analyzed (Participants) | 32 | 21 | 53 | 61 | 28
  Calcium (mmol/L): >1.1×ULN | 0 | 0 | 1 | 0 | 0
  Calcium (mmol/L): <0.9×LLN: number analyzed (Participants) | 32 | 21 | 53 | 61 | 28
  Calcium (mmol/L): <0.9×LLN | 1 | 0 | 0 | 0 | 0
  Chloride (mmol/L): <0.9×LLN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Chloride (mmol/L): <0.9×LLN | 0 | 0 | 1 | 0 | 0
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN: number analyzed (Participants) | 34 | 22 | 52 | 55 | 27
  Cholesterol, Total, Fasting (mmol/L): >1.6×ULN | 1 | 0 | 1 | 1 | 0
  Creatinine [micromoles(μmol)/L]: >1.3×ULN: number analyzed (Participants) | 29 | 20 | 50 | 57 | 26
  Creatinine [micromoles(μmol)/L]: >1.3×ULN | 0 | 3 | 5 | 7 | 3
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN: number analyzed (Participants) | 33 | 21 | 50 | 53 | 27
  Glucose-Chemistry, Fasting (mmol/L): >2.5×ULN | 5 | 2 | 12 | 7 | 4
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN: number analyzed (Participants) | 33 | 21 | 50 | 53 | 27
  Glucose-Chemistry, Fasting (mmol/L): <0.9×LLN | 0 | 2 | 4 | 2 | 0
  Glycohemoglobin A1C (%): Increase of >=0.5%: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Glycohemoglobin A1C (%): Increase of >=0.5% | 18 | 18 | 41 | 37 | 24
  Glycohemoglobin A1C (%): Increase of >=1%: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Glycohemoglobin A1C (%): Increase of >=1% | 18 | 18 | 41 | 36 | 24
  Phosphorus (mmol/L): >1.1×ULN: number analyzed (Participants) | 32 | 22 | 53 | 60 | 28
  Phosphorus (mmol/L): >1.1×ULN | 4 | 0 | 3 | 2 | 2
  Phosphorus (mmol/L): <0.9×LLN: number analyzed (Participants) | 32 | 22 | 53 | 60 | 28
  Phosphorus (mmol/L): <0.9×LLN | 0 | 0 | 0 | 2 | 0
  Potassium (mmol/L): <0.9×LLN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Potassium (mmol/L): <0.9×LLN | 0 | 0 | 1 | 0 | 0
  Protein, Total (g/L): <0.9×LLN: number analyzed (Participants) | 34 | 22 | 53 | 61 | 28
  Protein, Total (g/L): <0.9×LLN | 1 | 1 | 0 | 0 | 0
  Triglycerides, Fasting (mmol/L): >=3×ULN: number analyzed (Participants) | 33 | 22 | 49 | 54 | 27
  Triglycerides, Fasting (mmol/L): >=3×ULN | 2 | 2 | 1 | 1 | 3
  Uric Acid (Urate) (μmol/L): >1.1×ULN: number analyzed (Participants) | 21 | 18 | 43 | 47 | 19
  Uric Acid (Urate) (μmol/L): >1.1×ULN | 4 | 6 | 9 | 8 | 4
  Uric Acid (Urate) (μmol/L): <0.9×LLN: number analyzed (Participants) | 21 | 18 | 43 | 47 | 19
  Uric Acid (Urate) (μmol/L): <0.9×LLN | 1 | 1 | 3 | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Meaningful Trends for Vital Signs
Description: Vital Signs included assessments of heart rate, respiratory rate, systolic and diastolic blood pressure, and body temperature. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to approximately 22 months
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
Number analyzed (Participants) | 35 | 22 | 54 | 62 | 28
Participants | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Meaningful Trends in Electrocardiogram (ECG) Results
Description: A standard 12-lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Up to approximately 22 months
Population: Safety Population included all participants who received ≥1 administration of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
Number analyzed (Participants) | 35 | 22 | 54 | 62 | 28
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 22 months
Description: All-Cause Mortality is reported for all randomized participants. The Safety Population, all participants who received ≥1 administration of study treatment, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Relamorelin/Relamorelin/Relamorelin | Relamorelin/Placebo/Relamorelin | Placebo/Relamorelin/Relamorelin | Relamorelin/Relamorelin | Placebo/Relamorelin
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/22 | 0/54 | 0/63 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/35 | 3/22 | 7/54 | 2/62 | 0/28
Other Adverse Events (participants affected / at risk) | 10/35 | 6/22 | 15/54 | 10/62 | 7/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Relamorelin/Relamorelin/Relamorelin (N=35) | Relamorelin/Placebo/Relamorelin (N=22) | Placebo/Relamorelin/Relamorelin (N=54) | Relamorelin/Relamorelin (N=62) | Placebo/Relamorelin (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 2 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 1 | 0 | 0
Spinal claudication (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Thalamic infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Relamorelin/Relamorelin/Relamorelin (N=35) | Relamorelin/Placebo/Relamorelin (N=22) | Placebo/Relamorelin/Relamorelin (N=54) | Relamorelin/Relamorelin (N=62) | Placebo/Relamorelin (N=28)
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 2 | 5 | 3
Urinary tract infection (Infections and infestations) | 2 | 3 | 2 | 0 | 1
Vulvovaginal mycotic infection (Infections and infestations) | 0/26 | 1/14 | 0/38 | 0/45 | 1/22 — Number at risk is based on the female population.
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2 | 2 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 0 | 2
Headache (Nervous system disorders) | 1 | 0 | 4 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03786380/Prot_002.pdf
  • Statistical Analysis Plan (2020-09-30): https://cdn.clinicaltrials.gov/large-docs/80/NCT03786380/SAP_001.pdf